CLINICAL TRIAL: NCT02885142
Title: Early Rectal Cancer: Endoscopic Submucosal Dissection or Transanal Endoscopic Microsurgery?
Acronym: MUCEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties to recruit all the patients
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-33; 2016-A01363-48 (Other: Ansm)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transanal endoscopic microsurgery group (Experimental)
  Interventions: Procedure: Local excision for early rectal cancer
- endoscopic submucosal dissection group (Active Comparator)
  Interventions: Procedure: Local excision for early rectal cancer

INTERVENTIONS:
Procedure: Local excision for early rectal cancer

SUMMARY:
Local excision for early rectal cancer has proven its feasibility and oncological safety. Indeed, lymph node invasion does not exceed 1% and 10% in pT1sm1 and pT1sm2 rectal carcinomas respectively. Two procedures are currently performed in these early cancers as well as in preneoplastic lesions. Transanal endoscopic microsurgery (TEM), which has proven its superiority over traditional transanal excision, is a surgical approach associated with a 92% R0 excision rate, a survival comparable to radical anterior resection and a low morbidity. It consists of a full-thickness excision. The second procedure is a recently introduced technique: the endoscopic submucosal dissection (ESD), which encompasses only the mucosa and submucosa. ESD enables endoscopists to achieve higher en bloc resection rates than standard mucosectomy and is associated with a 88% R0 resection rate, which decreases to 65% in the subgroup of European series. Though very promising, the role of ESD remains controversial in malignant lesions with few published reports. There are therefore 2 different techniques with 2 different dissections (full-thickness vs. submucosal) to achieve the same oncological treatment. So far, only one retrospective single-center study including 63 patients has compared TEM and ESD in early rectal cancer without finding any difference between the 2 procedures, and there are no other available studies comparing TEM and ESD for any type of colorectal tumor. The aim of the present research is to compare ESD with TEM for early rectal cancer and rectal adenomas for short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with an ERT (i.e. rectal adenoma or rectal carcinoma Tis or staged usT1N0 on endorectal ultrasound) that can be alternately resectable by TEM or ESD
* Histology proved by a preoperative biopsy

Exclusion Criteria:

* " Palliative " excision T2/3/4 or N+
* Preoperative radiochemotherapy (down-staging)
* Metastatic cancer
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2016-11; Primary Completion 2020-06-11 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Number of complete excision for TEM compare to number of complete excision for ESD in rectal carcinomas staged usT1N0 and rectal adenomas. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Laura BEYER, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beyer-Berjot L, Delettrez C, Jacques J, Rouanet P, Chaussade S, Lefevre JH, Chabrun E, Koch S, Tuech JJ, Bridoux V, Rullier E, Denost Q, Panis Y, Maggiori L, Benoist S, Brouquet A, Barthet M, Gonzalez JM, Cotte E, Arquilliere J, Jafari M, Meurette G, Poincloux L, Zerbib P, Regimbeau JM, Sabbagh C, Prudhomme M, Legros R, Berdah S, Dervaux B, Boucekine M, Denies F, Rivory J, Baumstarck K, Pioche M, Lepilliez V. TEM OR ESD IN EARLY RECTAL TUMORS: A CLINICAL & COST-EFFECTIVENESS ANALYSIS. Gastroenterology. 2026 Jan 29:S0016-5085(26)00029-6. doi: 10.1053/j.gastro.2026.01.006. Online ahead of print. PMID 41620037